CLINICAL TRIAL: NCT03535714
Title: MANTR-a: Evaluation of a Therapeutic Intervention for Adolescents and Young Adults With Anorexia Nervosa
Brief Title: Maudsley Model of Anorexia Nervosa Treatment for Adolescents and Young Adults (MANTR-a)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: Pharmig - Gesundheitsziele aus dem Rahmen-Pharmavertrag (Other)
Responsible Party: Principal Investigator, Dr. Andreas Karwautz, Univ. Prof. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FA765A0306
Record Dates: First submitted 2018-03-28; First posted 2018-05-24 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Anorexia Nervosa; Anorexia
Keywords: Treatment; Psychotherapy; Young Adult; Adolescence
MeSH Terms: conditions — Anorexia Nervosa; Anorexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MANTR-a group (Active Comparator): Patients who are in the MANTR-a group attend the MANTR-a treatment program, which consists of 20 once-weekly therapy sessions. Caregivers can be invited to 2 sessions. After 20 weeks, therapy continues with four monthly booster-sessions. In sum, each patient (whose bodyweight is above the 3rd BMI percentile) can attend 24 therapy sessions. In patients whose bodyweight is below the 3rd BMI percentile treatment will be extended to 30 once-weekly and 4 monthly booster sessions. Besides therapy the patients are in nutritional consultation by a dietician and under regular medical care to monitor the physical health and weight gain.
  Patients who who have already an existing psychotherapy are attached to the control group.
  Interventions: Behavioral: MANTR-a treatment
- control group (No Intervention): Patients of the control group receive treatment as usual (TAU). It consists of medical care and monitoring, psychotherapy in a single or family setting, parents counselling and dietetics.

INTERVENTIONS:
Behavioral: MANTR-a treatment — MANTR-a treatment
  Arms: MANTR-a group

SUMMARY:
The aim of this study is to test effectiveness of a new treatment program for adolescents and young adults within the age of 14-21 suffering from AN (MANTR-a) compared to treatment as usual (TAU).

DETAILED DESCRIPTION:
Anorexia nervosa (AN) is a serious mental illness which leads untreated to aggravation of symptomatology and chronification. Among all mental illnesses, AN has the highest mortality rate, which is about 5.1 per 1000 people per year. High drop-out rates (up to 40%) or small treatment motivation constrains treatment success. Since the onset of AN is mainly in adolescence, it is important to start with therapy as early as possible and establish an effective single-setting treatment program for this age group to prevent chronification.

MANTR-a (Maudsley model of anorexia nervosa treatment for adolescents) is an innovative, theory-based, tailored treatment program which combines a cognitive behavioural approach with motivational interviewing. The main focus of the treatment program is the transformation maintaining factors of AN, like personality aspects, pro-anorexic beliefs, emotion regulation strategies, thinking styles and obstructive behaviour from caregivers.

The aim of this study is the examination ot the effectiveness of the MANTR-a treatment program for adolescents and young adults. Therefore we compare MANTR-a (intervention group) with treatment as usual (control group). Assessments will be conducted before treatment (T0, baseline), after six months (T1), after 12 months (T2) and after 18 months (T3, follow-up) via questionnaires, interviews and neuropsychological measurements. Process evaluation takes place after every session. Each group consists of female adolescents and young adults within the age of 14-21 suffering from AN (ICD-10: F50.0, F50.1), resulting in an overall sample size of 100.

The long-term goal of the study is to provide an evidence-based outpatient treatment for children and adolescents with AN in order to prevent a chronic course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of anorexia nervosa (F50.0) or atypical anorexia nervosa (F50.1).

Exclusion Criteria:

* life-threatening AN requiring immediate inpatient treatment as defined by NICE (2017)
* insufficient cognitive ability
* insufficient knowledge of German language to understand the treatment
* severe mental or physical illness that needs treatment on its own (e.g. psychosis)
* substance abuse
* pregnancy

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Increase of BMI | 12 months
  Weight and height will be assessed and combined to report BMI in kg/m^2
Improvement of eating disorder symptomatology based on professional's rating | 12 months
  Professionals use a structured clinical interview ("Eating Disorder Examination - EDE") to rate severity of eating disorder symptomatology
Improvement of eating disorder symptomatology based on patient's self-rating | 12 months
  "Eating Disorder Inventory-2 (EDI-2)" is used to assess eating disorder symptomatology from a patients's view

SECONDARY OUTCOMES:
Increase of BMI | 6 months, 18 months
  Weight and height will be assessed and combined to report BMI in kg/m^2
Improvement of eating disorder symptomatology based on professional's rating | 6 months, 18 months
  Professionals use a structured clinical interview ("Eating Disorder Examination - EDE") to rate severity of eating disorder symptomatology
Improvement of eating disorder symptomatology based on patient's self-rating | 6 months, 18 months
  "Eating Disorder Inventory-2 (EDI-2)" is used to assess eating disorder symptomatology from a patients's view
Group differences: increase of BMI | 6 months, 12 months, 18 months
  Group differences are calculated based on BMI (weight and height will be assessed and combined to report BMI in kg/m^2)
Group differences: improvement of eating disorder symptomatology based on professional's rating | 6 months, 12 months, 18 months
  Group differences are calculated based on professional's rating in a structured clinical interview ("Eating Disorder Examination - EDE)"
Group differences: improvement of eating disorder symptomatology based on patient's self-rating | 6 months, 12 months, 18 months
  Group differences are calculated based on a patient's self-rating questionnaire ("Eating Disorder Inventory-2")
Improvement of comorbid symptomatology based on professional's rating | 6 months, 12 months, 18 months
  Professionals use a structured clinical interview ("Diagnostisches Interview bei psychischen Störungen im Kindes- und Jugendalter") to rate severity of comorbid symptomatology
Reduction of anxiety | 6 months, 12 months, 18 months
  "State-Trait-Angstinventar (STAI X1, STAI X2)" is used to assess severity of anxiety from a patients's view
Reduction of depression | 6 months, 12 months, 18 months
  "Beck Depressionsinventar (BDI-II)" is used to assess severity of depression from a patients's view
Reduction of obsessive-compulsive symptomatology | 6 months, 12 months, 18 months
  "Zwangsinventar (OCI-R)" is used to assess severity of obsessive-compulsive symptomatology from a patients's view
Increase of cognitive flexibility | 12 months
  Cognitive flexibility is measured with "Computergestütztes Kartensortierverfahren (CKV)"
Increase of central coherence | 12 months
  Central coherence is measured with "Rey-Osterrieth Complex Figure Test (ROCF)"
Increase of emotion recognition | 12 months
  Emotion recognition is measured with "Frankfurter Program to test and to teach the recognition of facial affect (FEFA-2)"
Influence of motivation of change | 12 months
  Motivation of change is measured with "Anorexia nervosa Stages of Change Questionnaire (ANSOCQ)"
Quality of life (group differences, improvement over time) | 6 months, 12 months, 18 months
  Quality of Life is measured with "Lebensqualität von Kindern und Jugendlichen (ILK)"
Influence of therapeutic relationship | 6 months, 12 months
  Therapeutic relationship is measured with "Fragebogen zur therapeutischen Beziehung für Kinder und Jugendliche (FTB-KJ)"
Influence of treatment contentment | 6 months, 12 months
  Treatment contentment is measured with "Fragebogen zur Beurteilung der Behandlung (FBB)"
Changes in personality | 12 months
  Changes in personality are measured with "Junior Temperament und Charakter Inventar (JTCI 12-18R)"

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karwautz, Univ.-Prof., Study Director — Medical University of Vienna; Gudrun Wagner, Ass.-Prof., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Dep. of Child and Adolescent Psychiatry, Vienna, Austria

REFERENCES:
- [Background] Arcelus J, Mitchell AJ, Wales J, Nielsen S. Mortality rates in patients with anorexia nervosa and other eating disorders. A meta-analysis of 36 studies. Arch Gen Psychiatry. 2011 Jul;68(7):724-31. doi: 10.1001/archgenpsychiatry.2011.74. PMID 21727255
- [Background] Dejong H, Broadbent H, Schmidt U. A systematic review of dropout from treatment in outpatients with anorexia nervosa. Int J Eat Disord. 2012 Jul;45(5):635-47. doi: 10.1002/eat.20956. Epub 2011 Aug 30. PMID 22684990
- [Background] Schmidt U, Treasure J. Anorexia nervosa: valued and visible. A cognitive-interpersonal maintenance model and its implications for research and practice. Br J Clin Psychol. 2006 Sep;45(Pt 3):343-66. doi: 10.1348/014466505x53902. PMID 17147101
- [Background] Treasure J, Schmidt U. The cognitive-interpersonal maintenance model of anorexia nervosa revisited: a summary of the evidence for cognitive, socio-emotional and interpersonal predisposing and perpetuating factors. J Eat Disord. 2013 Apr 15;1:13. doi: 10.1186/2050-2974-1-13. eCollection 2013. PMID 24999394
- [Derived] Wittek T, Zeiler M, Truttmann S, Philipp J, Kahlenberg L, Schneider A, Kopp K, Krauss H, Auer-Welsbach E, Koubek D, Ohmann S, Werneck-Rohrer S, Sackl-Pammer P, Laczkovics C, Mitterer M, Schmidt U, Karwautz A, Wagner G. The Maudsley model of anorexia nervosa treatment for adolescents and emerging adults: A multi-centre cohort study. Eur Eat Disord Rev. 2025 Nov;33(6):1117-1132. doi: 10.1002/erv.2996. Epub 2023 Jun 11. PMID 37302134
- [Derived] Wittek T, Truttmann S, Zeiler M, Philipp J, Auer-Welsbach E, Koubek D, Ohmann S, Werneck-Rohrer S, Sackl-Pammer P, Schofbeck G, Mairhofer D, Kahlenberg L, Schmidt U, Karwautz AFK, Wagner G. The Maudsley model of anorexia nervosa treatment for adolescents and young adults (MANTRa): a study protocol for a multi-center cohort study. J Eat Disord. 2021 Mar 8;9(1):33. doi: 10.1186/s40337-021-00387-8. PMID 33685522